CLINICAL TRIAL: NCT03542123
Title: Cardiac Output Autonomic Stimulation Therapy for Heart Failure - Hemodynamic Effects
Acronym: COAST-HF FX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuroTronik Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 700003-02
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure Acute; Heart Failure
Keywords: Electrical Stimulation Therapy; Electrodes; Parasympathetic Nervous System; Sympathetic Fibers, Post Ganglionic; Congestive Heart Failure; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeuroTronik CANS Therapy® System (Experimental)
  Interventions: Device: NeuroTronik CANS Therapy® System

INTERVENTIONS:
Device: NeuroTronik CANS Therapy® System — The NeuroTronik CANS Therapy® System is a percutaneous, catheter-based, bedside electrical stimulation system. The System consists of the single-use, disposable NeuroCatheter™ and NeuroCatheter™ Placement Kit, along with the reusable, bedside NeuroModulator™ Development System, and the NeuroTronik CANS Therapy™ Cable.

SUMMARY:
A single-arm study to observe NeuroTronik Cardiac Autonomic Nerve Stimulation (CANS) Therapy System hemodynamic and other physiologic effects.

ELIGIBILITY:
Inclusion Criteria:

* Normal sinus rhythm by ECG
* Men and women 21-75 years old
* Patients with stable symptomatic heart failure, New York Heart Association (NYHA) class II, III, or IV.

Exclusion Criteria:

* Systolic Blood Pressure < 90 mmHg or > 160 mmHg
* Current amiodarone therapy or any other antiarrhythmic therapy
* Coronary artery bypass graft surgery or percutaneous coronary intervention within prior 1 month
* Enzyme-positive MI within prior 1 month
* Patients who have been hospitalized for heart failure and who required the use of HF IV therapy within 30 days before enrollment (measured from release)
* History of recent severe ventricular arrhythmias
* Pre-existing carotid artery or cerebral disease
* Patients with hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g. amyloidosis, sarcoidosis)
* Patients with prior vagalotomy
* Patients with current or prior vagal nerve stimulators
* Subjects with narrow angle glaucoma
* Renal failure - on dialysis or serum creatinine > 2.0 mg/dl
* Hepatic failure - bilirubin, SGOT, or SGPT > 4X upper limit of normal
* Patients with a life expectance < 12 months per physician judgment
* Women who are pregnant
* Allergy to fentanyl, midazolam, propofol, eggs, egg products, soybeans, or soy products
* Subjects unwilling or unable to provide consent for the protocol

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricular pressure and volume | One hour

SECONDARY OUTCOMES:
Heart rate | One hour

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay